CLINICAL TRIAL: NCT02116504
Title: Multi-center Prospective European Cohort Study in Patients With Rheumatoid Arthritis or Juvenile Idiopathic Arthritis Planned to be Treated Independently of the Present Study, With the First Line of Adalimumab, Etanercept, Infliximab Therapy or With Rituximab or Tocilizumab (After Anti-Tumor Necrosis Factor Therapy or Another Biotherapy or in First Line)
Brief Title: Anti-Biopharmaceutical Immunization: Prediction and Analysis of Clinical Relevance to Minimize the Risk of Immunization in Rheumatoid Arthritis Patients or Juvenile Idiopathic Arthritis Patients
Acronym: ABI-RA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Leiden University Medical Center (Other); University College London (UCL) Cancer Institute (Other); University of Florence (Other); Pediatric Rheumatology International Trials Organization (Other); Istituto Giannina Gaslini (Other); GlaxoSmithKline (Industry); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ABI-RA-P01; 2013-A01268-37 (Other: ANSM)
Record Dates: First submitted 2014-04-03; First posted 2014-04-17 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis; Juvenile Idiopathic Arthritis
Keywords: Rheumatoid arthritis; Juvenile Idiopathic Arthritis; Biopharmaceutical; Immunogenicity; Anti-Drug Antibody; Prediction
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Global population (Other): All included patients :
  Sampling of blood
  Interventions: Procedure: Sampling of blood

INTERVENTIONS:
Procedure: Sampling of blood — Sampling of blood for dosage of antibodies

SUMMARY:
One of the main potential causes of these failures of BP therapy response is the development of Anti-drug Anti-body (ADAb) in some patients. ADAb may decrease the efficacy of BPs by neutralizing them or modifying their clearance and they may be associated with BP-specific hypersensitivity reactions. The prediction, prevention and cure of anti-drug (AD) immunization are thus major goals in BP development. This prospective study (ABI-RA) will assess the occurrence of ADAb using standardized and validated assay(s) and also cellular, genetic and molecular parameters in RA/JIA patients treated with adalimumab, etanercept, infliximab and rituximab or tocilizumab, to address the mechanism of immunogenicity. Patient-related factors that might predispose an individual to an immune response will be taken into account: underlying disease, genetic background, immune status, including immunomodulating therapy and dosing schedule.

DETAILED DESCRIPTION:
The ABIRISK (Anti-biopharmaceutical Immunization: Prediction and analysis of clinical relevance to minimize the risk) consortium, within the IMI (Innovative Medicines Initiative), is a Public Private Partnership between pharmaceutical companies, academic institutions and clinical centers. The ABIRISK aims are to better analyze and predict the phenomenon of immunogenicity in order to reduce its occurrence. One of the main objectives of ABIRISK is to set up prospective cohort (ABI-RA) of patients with rheumatoid arthritis (RA) or juvenile idiopathic arthritis (JIA) to provide, using an integrated approach, new tools for being able to detect earlier and even before the beginning of the therapy, immunization to biopharmaceutical (BP). The introduction of BP has been a critical step forward in care for RA/JIA and 9 BP are now licensed for the treatment of RA/JIA. In spite of this progress, failure of response to BP is frequent and in most of the registries, less than 50 % of patients are still on drug at 5 years. These failures may be primary failures or secondary failures. The fact is that the low level of responses becomes insufficient compared to the expectations. One of the main potential causes of these failures of BP therapy response is the development of Anti-drug Anti-body (ADAb) in some patients. ADAb may decrease the efficacy of BPs by neutralizing them or modifying their clearance and they may be associated with BP-specific hypersensitivity reactions. The prediction, prevention and cure of anti-drug (AD) immunization are thus major goals in BP development. This prospective study (ABI-RA) will assess the occurrence of ADAb using standardized and validated assay(s) and also cellular, genetic and molecular parameters in RA/JIA patients treated with adalimumab, etanercept, infliximab and rituximab or tocilizumab, to address the mechanism of immunogenicity. Patient-related factors that might predispose an individual to an immune response will be taken into account: underlying disease, genetic background, immune status, including immunomodulating therapy and dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of more than 18 years old diagnosed with RA according to 2010 ACR/EULAR criteria Or Male and female patients Age > 2 years and <18 years, diagnosed with JIA according to the Internal League Against Rheumatism (ILAR) classification criteria.
* Patient for whom the Treating Physician has decided to prescribe in the usual manner in accordance with the terms of the marketing authorization and independently from entry into this study:
* etanercept, adalimumab, infliximab, infliximab Biosimilar, rituximab OR tocilizumab in first line or after failure with other biotherapy. In case of previous rituximab, inclusion may be possible at least 6 months after the last rituximab infusion therapy or,
* Subcutaneous form of Tocilizumab, either as first line or after switch from infusion tocilizumab form is allowed.
* Having given written informed consent prior to undertaking any study-related procedures. For JIA patients, written informed consent signed by parents or legal representative and assent of the minor child
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research

Exclusion Criteria:

* Under any administrative or legal supervision.
* Patients having previously anti-TNF if they are going to receive another anti-TNF therapy
* Patients having previously received rituximab in the past 6 months.
* Conditions/situations such as:

  * Patients with conditions/concomitant diseases making them non evaluable for the primary endpoint
  * Impossibility to meet specific protocol requirements (e.g. blood sampling)
  * Patient is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
  * Uncooperative or any condition that could make the patient potentially non-compliant to the study procedures
* Pregnant or breast-feeding women

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Immunization against the Biopharmaceutical defined by the presence of ADAb within the first 12 months (or W52) | 52 weeks

SECONDARY OUTCOMES:
Quantification of ADAb | at Week 0
Quantification of ADAb | at Week 4
Quantification of ADAb | at Week 12
Quantification of ADAb | at Week 26
Quantification of ADAb | at Week 52
Quantification of ADAb | at Week 64
Quantification of ADAb | at Week 78
Clinical response and remission | at Week 4
  European League Against Rheumatism (EULAR) response
Clinical response and remission | at Week 12
  European League Against Rheumatism (EULAR) response
Clinical response and remission | at Week 26
  European League Against Rheumatism (EULAR) response
Clinical response and remission | at Week 52
  European League Against Rheumatism (EULAR) response
Clinical response and remission | at Week 64
  European League Against Rheumatism (EULAR) response
Clinical response and remission | at Week 78
  European League Against Rheumatism (EULAR) response
ADAb-associated adverse clinical events at any time point | Until Week 78
Drug levels | Until week 78
  Concentration in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paoletti A, Ly B, Bitoun S, Nocturne G, Riviere E, Manson JJ, Matucci A, Pallardy M, De Vries N, Mariette X. Restoration of Default Blood Monocyte-Derived Macrophage Polarization With Adalimumab But Not Etanercept in Rheumatoid Arthritis. Front Immunol. 2022 Feb 23;13:832117. doi: 10.3389/fimmu.2022.832117. eCollection 2022. PMID 35281074
- [Derived] Duhaze J, Caubet M, Hassler S, Bachelet D, Allez M, Deisenhammer F, Fogdell-Hahn A, Gleizes A, Hacein-Bey-Abina S, Mariette X, Pallardy M, Broet P; ABIRISK Consortium. Assessing the effect of genetic markers on drug immunogenicity from a mechanistic model-based approach. BMC Med Res Methodol. 2020 Mar 20;20(1):69. doi: 10.1186/s12874-020-00941-z. PMID 32192445
- [Derived] Bitoun S, Nocturne G, Ly B, Krzysiek R, Roques P, Pruvost A, Paoletti A, Pascaud J, Donnes P, Florence K, Gleizes A, Hincelin-Mery A, Allez M, Hacein-Bey-Abina S, Mackay F, Pallardy M, Le Grand R, Mariette X. Methotrexate and BAFF interaction prevents immunization against TNF inhibitors. Ann Rheum Dis. 2018 Oct;77(10):1463-1470. doi: 10.1136/annrheumdis-2018-213403. Epub 2018 Jun 23. PMID 29936438